CLINICAL TRIAL: NCT01311752
Title: Study of Human Papillomavirus Related Genital Pathology Among HIV Positive
Brief Title: Study of Human Papillomavirus Related Genital Pathology Among HIV Positive Women
Acronym: ANRS CO17
Status: Completed | Type: Observational
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Virology study Heather A Cubie Catherine Moore Edinburg United Kingdom (Unknown); Anatomopathology study Christine Bergeron Laboratoire Pasteur Cerba Cergy Pontoise France (Unknown); Paris, Isabelle Cartier, M.D. (Individual); Immunology study Guislaine Carcelain Groupe Hospitalier Pitié Salpétrière Paris (Unknown); Surgery study Hervé Foulot Cochin Paris (Unknown)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Other Study IDs: 2007-A00703-50
Record Dates: First submitted 2010-07-16; First posted 2011-03-09 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: HIV Infections
Keywords: human papillomavirus; follow up
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: surgical management of high grade lesions — Clinical, pathological and biological, data at diagnosis and during follow-up will be collected.
  Surgical sample will be collected to study human papillomavirus related genital pathology.

SUMMARY:
This study is a Multicentre cohort study with inclusion throughout the full duration of the study.

The primary objective is the study of human papillomavirus related genital pathology in HIV positive women.

The secondary objective are:

1. To study the characteristics of HPV infection and related disease in the context of long term HAART and HIV infection ;
2. To study the characteristics of atypical cells of uncertain significance detected in Pap smears, whose prevalence has dramatically increased in the last years;
3. To describe cervical cancers observed in the cohort
4. To study the evolution of recurrent high-grade lesions after surgery
5. To describe the evolution of vaginal lesions developed after hysterectomy for high-grade lesions ;
6. To describe the specific aspects of surgery for the treatment of cervical lesions according to the specific localization in the endocervix in HIV-positive women ;
7. To study the in situ T cell HPV specific response in cervical lesions and the relationship between virological and clinical parameters, host immune status and natural history of lesions ;
8. To initiate a prospective study on anal HPV infection and related disease among women infected with HIV.
9. To initiate a study on therapeutic and/or prophylactic HPV vaccines in the context of immunosuppression and a high rate of HPV infection ;

DETAILED DESCRIPTION:
Data were be collected into evaluate:

* Analysis of prognostic factors (CD4, antiviral therapy) of cervical lesions, using Cox models.
* Estimation of rates of Incidence of high grade lesions, of recurrence after surgical treatments using Kaplan Meier tests.
* Logistic regression analysis for the study of factors associated with complete excision after surgical treatment.
* SIR (standardised incidence rate) evaluation for cervical cancer

Study procedures are Annual follow-up in case of normal Pap smear, biannual follow-up in case of cervical lesions. Surgical management of High grade lesions.

ELIGIBILITY:
Inclusion Criteria:

* women > 18 years old
* attending outpatient gynecology consultation
* HIV positive
* with written informed consent
* on social security

Exclusion Criteria:

* unaffiliated to the social healthy security french system

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 676 (Actual)
Dates: Start 2007-11; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Heard, MD, Principal Investigator — Unité biologie de la reproduction, GH Pitié Salpétrière; Manuella Bonmarchand, Principal Investigator — Service Médecine Interne La Pitié Salpétrière; Roland Tubiana, Principal Investigator — Service maladies infectieuses La Pitié Salpétrière; Ana Canestri, Principal Investigator — Service maladies infectieuses La Pitié Salpétrière; Catherine Creen Hebert, Principal Investigator — Service Gynécologie-obstétrique Louis Mourier; Laurent Mandelbrot, Principal Investigator — Service Gynécologie Louis Mourier; Francoise Meier, Principal Investigator — Service Gynécologie Louis Mourier; Elisabeth Foucher, Principal Investigator — Service Gynécologie Louis Mourier; Marie Jeanne Ducassou, Principal Investigator — Hopital de jour CISIH Marseille; Isabelle Poizot Martin, Principal Investigator — Hôpital de jour CISIH Marseille; Bénédicte Lefèvre, Principal Investigator — Service des maladies infectieuses St Antoine; Bruno Carbonne, Principal Investigator — Service Gynécologie St Antoine; Dahlia Torchin, Principal Investigator — Service Gynécologie St Antoine; Anne Isabelle Richet, Principal Investigator — Service Gynécologie St Antoine; Jean Paul Viard, Principal Investigator — centre de diagnostic et thérapeutique Hopital Hotel Dieu; Christine Rousset Jablonski, Principal Investigator — Service Gynécologie Obstétrique Hopital Hotel Dieu

REFERENCES:
- See also: Related Info — http://anrs.fr